CLINICAL TRIAL: NCT06637956
Title: The Effect of Intranasally Administered Nitroglycerin on Hemodynamic Response to Laryngoscopy and Intubation Among Patients Undergoing Coronary Artery Bypass Grafting (CABG) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC_Lahore
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Intranasal; nitroglycerin; hemodynamic response; larayngoscopy; intubation; coronary artery bypass grafting
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NTG (Experimental): Received a mg nitroglycerin intranasally two minutes prior to laryngoscopy and intubation
  Interventions: Drug: Nitroglycerin (NTG)
- Control (No Intervention): Control group did not receive nitroglycerine prior to laryngoscopy and intubation

INTERVENTIONS:
Drug: Nitroglycerin (NTG) — Received 1 mg of nitroglycerin intranasally two minutes prior to laryngoscopy and intubation
  Arms: NTG

SUMMARY:
Numerous preventive medications have been used to lessen the cardiovascular response to laryngoscopy and intubation. Though some advantages have been noted, most of these treatments have not been found to be completely satisfying. However, nitroglycerin is the most widely utilized medicine due to its fast effect, short half-life, and absence of sedative qualities.

DETAILED DESCRIPTION:
The circulatory system under compromise is less resilient to the effects of general anaesthesia. Inducing anaesthesia is a crucial step for cardiac patients because their impaired circulatory systems are less tolerant to depression. During coronary artery bypass grafting surgery, the primary objective of general anesthesia is to reduce sympathetic response to uncomfortable stimuli, including laryngoscopy, intubation, skin incision, sternal splitting, and spreading. A rise in blood pressure is one of the hemodynamic reactions that is typically associated with tracheal intubation and laryngoscopy. The impact of intra nasally delivered nitroglycerin on blood pressure response to laryngoscopy and intubation in patients having non-cardiac surgery is currently contentious; however, this study focus on coronary artery bypass grafting surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Patients undergoing coronary artery bypass grafting surgery.
* Patients aged 35-60 years.
* Ejection Fraction between 50-60%.
* American Society of Anesthesiologists Classification 3-4.

Exclusion Criteria:

* Known hypersensitivity to nitroglycerin.
* Anticipated difficult airway.
* Emergency surgery.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mean aterial pressure | 5 minutes post intubation
  Mean arterial pressure was measured prior to and after intubation
Heart rate | 5 minutes post intubation
  Heart rate was measure prior to and after intubation
Systolic blood pressure | 5 minutes post intubation
  Systolic blood pressure was measure prior to and after itubation
Diastolic blood pressure | 5 minutes post intubation
  Diastolic blood pressure was measure prior to and after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Shehryar Ahmed, MS, Principal Investigator — Department of anesthesia Rashid Latif Medical college, Lahore, Pakistan; Syed Shakeel Ahmed, FCPS, Principal Investigator — Department of Anesthesia, Shahida Islam Teaching Hospital, Lodhran, Pakistan
Locations (1):
- Department of Anesthesia, Rashid Latif Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No